CLINICAL TRIAL: NCT07037576
Title: Efficacy and Safety of Prepectoral Prosthesis Immediate One-Stage Breast Reconstruction Versus Two-Stage Expander/Prosthesis Reconstruction in Postoperative Adjuvant Radiotherapy Breast Cancer Patients: A Prospective, Single-Center, Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2025-034
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer Patients
Keywords: Breast cancer; Breast reconstruction surgery; Radiotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Immediate One-Stage Prepectoral Prosthetic Breast Reconstruction Cohort: Patients undergoing nipple-sparing mastectomy (NSM) or skin-sparing mastectomy (SSM) with immediate prepectoral prosthetic breast reconstruction are eligible for inclusion, regardless of mesh use (with or without mesh). Approaches including open, endoscopic, or robotic techniques are acceptable, provided that adjuvant radiotherapy is administered after permanent implant placement.
  Interventions: Procedure: Breast Reconstruction Surgery
- Delayed-Immediate Two-Stage Expander/Implant Breast Reconstruction Cohort: Patients undergoing nipple-sparing mastectomy (NSM) or skin-sparing mastectomy (SSM) with two-stage expander/implant breast reconstruction are eligible, provided that: Expander placement may be either prepectoral or subpectoral, Mesh use is optional (with or without acellular dermal matrix), Radiotherapy is administered with the expander in situ, Permanent implant exchange is performed ≥6 months after completing radiotherapy, The implant exchange procedure permits any approach (open, endoscopic, or robotic) and any plane/mesh configuration (prepectoral/subpectoral, with/without mesh).
  Interventions: Procedure: Breast Reconstruction Surgery

INTERVENTIONS:
Procedure: Breast Reconstruction Surgery — Breast Reconstruction Surgery (either immediate one-stage prepectoral implant reconstruction or two-stage expander/implant reconstruction) with postoperative adjuvant radiotherapy
  Other Names: radiation

SUMMARY:
Prospective Evaluation of the Efficacy and Safety of Prepectoral Immediate One-Stage Prosthetic Breast Reconstruction Versus Two-Stage Expander/Prosthesis Reconstruction in Postoperative Adjuvant Radiotherapy Breast Cancer Patients

DETAILED DESCRIPTION:
This study is a prospective, double-cohort study. It plans to enroll more than 104 patients with cT1-3N0-3M0 breast cancer for immediate prepectoral muscle prosthesis reconstruction or two-step breast reconstruction with expander/prosthesis, and they will receive postoperative radiotherapy. Record the changes of BREAST-Q scores of the patients before and after the operation, as well as information such as postoperative complications and capsular contracture.

The primary endpoint was the BREAST-Q score at 12 months after the operation. The secondary endpoints included the success rate of breast reconstruction, surgical complications, cosmetic effects of the breast evaluated by doctors, the occurrence of capsular contracture, nipple and skin sensation, and tumor safety.

ELIGIBILITY:
Inclusion Criteria:

1. women aged 18 to 70；
2. Newly diagnosed breast cancer patients showing no evidence of distant metastasis on clinical examination and diagnostic workup；
3. adjuvant radiotherapy is required;
4. Patients scheduled to undergo nipple-sparing mastectomy (NSM) or skin-sparing mastectomy (SSM) with immediate prepectoral implant-based reconstruction (via open, endoscopic, or robotic approach) require adjuvant radiotherapy AFTER permanent implant placement; OR Patients scheduled for NSM/SSM with two-stage tissue expander/implant reconstruction (with expander placement in either submuscular or prepectoral plane) receive radiotherapy WITH the tissue expander in situ, followed by exchange for permanent implant ≥6 months post-radiotherapy (expander position: submuscular/prepectoral acceptable; surgical approach: open/endoscopic/robotic acceptable);
5. Patients are eligible regardless of whether mesh is used in the reconstruction surgery;
6. Patients with severe breast ptosis are eligible;
7. During the study observation period, lipofilling is permitted on the affected breast and symmetrization procedures on the contralateral breast in both cohorts;
8. ECOG performance status 0-1;
9. Patients receiving neoadjuvant chemotherapy (NACT) are eligible;
10. Bilateral breast reconstruction is permitted;
11. No smoking history OR smoking cessation ≥4 weeks prior to enrollment;
12. Investigator-confirmed protocol compliance capability;
13. Concurrent participation in other interventional/non-interventional trials is allowed if deemed non-interfering by the investigator;
14. Voluntarily participate and sign the informed consent form after comprehensive understanding.

Exclusion Criteria:

1. Stage IV (metastatic) breast cancer;
2. No prior radiotherapy post-mastectomy;
3. History of ipsilateral chest wall/axillary radiation therapy;
4. Immunodeficiency, poorly controlled diabetes (HbA1c >7%), or active tobacco use;
5. Inflammatory breast cancer (cT4d);
6. Autologous-based breast reconstruction or delayed reconstruction;
7. Severe cardiopulmonary/hepatic/renal comorbidities contraindicating surgery/radiotherapy (ASA class ≥III);
8. Psychiatric disorders precluding independent BREAST-Q completion;
9. Pregnancy or lactation;
10. Documented history of protocol non-adherence;
11. Life-limiting comorbidities interfering with treatment OR investigator-determined ineligibility.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Treatment-naïve women with unilateral primary breast cancer (clinical stage cT1-3N0-3M0) scheduled for immediate prepectoral direct-to-implant reconstruction OR tissue expander/implant two-stage reconstruction, followed by adjuvant radiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
BREAST-Q (Breast Reconstruction Module) Scores | Preoperatively and at 1 Year Postoperatively
  This trial collects patient-reported outcomes through four domains of the BREAST-Q Breast Reconstruction Module: Satisfaction with Breasts, Psychosocial Well-being, Physical Well-being, Sexual Well-being. Scores are assessed preoperatively and at 12 months postoperatively. The BREAST-Q score at 12 months post-surgery serves as the primary endpoint.

SECONDARY OUTCOMES:
Breast Reconstruction Failure Rate | 1 Year Postoperatively
  Breast Reconstruction Failure Rate: Defined as the proportion of patients requiring implant removal due to complications among all patients undergoing breast reconstruction. Implant Removal Due to Complications: Refers to explantation occurring within 12 months postoperatively attributed to any of the following surgery-related complications: Hematoma, Seroma, Flap necrosis, Nipple-areolar complex (NAC) necrosis, Surgical site infection, Wound dehiscence, Implant exposure, Baker grade III/IV capsular contracture, Implant malposition/displacement. Exclusion Criterion: Implant removals requested by patients without objective surgery-related complications (i.e., subjectively motivated explantations) must be documented separately and excluded from failure rate calculations.
Complication Profile: | 1 Year Postoperatively
  Includes but not limited to: Hematoma, Poor Wound Healing, Flap Necrosis, Surgical Site Infection, Wound Dehiscence, Fat Grafting-Associated Complications. All complications must be graded according to the Clavien-Dindo Classification System, then systematically assessed and documented.
Physician-Assessed Aesthetic Outcome | 1 Year Postoperatively
  Evaluated by surgeons independent of the operating team using the Harris Scale to grade the aesthetic outcome of the reconstructed breast based on standardized patient photographs.
Capsular Contracture Assessment | 1 Year Postoperatively
  Evaluated using the Baker Classification System (Spear & Baker, 1995).
Nipple and Skin Sensation Assessment | 1 Year Postoperatively
  Tactile sensation is evaluated using the Semmes-Weinstein Monofilament Examination (SWME).
Oncological Safety Endpoints: Disease-Free Survival (DFS) and Overall Survival (OS). | 5 Year Postoperatively
  DFS: Time interval from the date of surgery to the occurrence of any recurrence (local/regional/distant metastasis), new primary breast cancer, or death from any cause, whichever occurs first. Patients without events are censored at the last documented disease-free follow-up.
  OS: Time interval from the date of surgery to death from any cause. Living patients are censored at the last confirmed survival follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: xiuchun chen, Study Director — Henan Cancer Hospital
Locations (1):
- Henan cacer hospital, Henan, Henan, China

REFERENCES:
- [Result] Kraenzlin F, Chopra K, Kokosis G, Venturi ML, Mesbahi A, Nahabedian MY. Revision Breast Reconstruction with Prepectoral Pocket Conversion of Submuscular Breast Implants. Plast Reconstr Surg. 2021 May 1;147(5):743e-748e. doi: 10.1097/PRS.0000000000007885. PMID 33890886
- [Result] Chatterjee A, Nahabedian MY, Gabriel A, Macarios D, Parekh M, Wang F, Griffin L, Sigalove S. Early assessment of post-surgical outcomes with pre-pectoral breast reconstruction: A literature review and meta-analysis. J Surg Oncol. 2018 May;117(6):1119-1130. doi: 10.1002/jso.24938. Epub 2018 Jan 18. PMID 29346711
- [Result] Li Y, Xu G, Yu N, Huang J, Long X. Prepectoral Versus Subpectoral Implant-Based Breast Reconstruction: A Meta-analysis. Ann Plast Surg. 2020 Oct;85(4):437-447. doi: 10.1097/SAP.0000000000002190. PMID 31913902
- [Result] Sigalove S. Prepectoral breast reconstruction and radiotherapy-a closer look. Gland Surg. 2019 Feb;8(1):67-74. doi: 10.21037/gs.2019.01.01. PMID 30842930
- [Result] Gabriel A, Maxwell GP. Prepectoral Breast Reconstruction in Challenging Patients. Plast Reconstr Surg. 2017 Dec;140(6S Prepectoral Breast Reconstruction):14S-21S. doi: 10.1097/PRS.0000000000004046. PMID 29166343
- [Result] Chopra S, Al-Ishaq Z, Vidya R. The Journey of Prepectoral Breast Reconstruction through Time. World J Plast Surg. 2021 May;10(2):3-13. doi: 10.29252/wjps.10.2.3. PMID 34307092
- [Result] Clemens MW, Kronowitz SJ. Acellular dermal matrix in irradiated tissue expander/implant-based breast reconstruction: evidence-based review. Plast Reconstr Surg. 2012 Nov;130(5 Suppl 2):27S-34S. doi: 10.1097/PRS.0b013e318265f690. PMID 23096982
- [Result] Kronowitz SJ, Hunt KK, Kuerer HM, Babiera G, McNeese MD, Buchholz TA, Strom EA, Robb GL. Delayed-immediate breast reconstruction. Plast Reconstr Surg. 2004 May;113(6):1617-28. doi: 10.1097/01.prs.0000117192.54945.88. PMID 15114121
- [Result] Sbitany H, Gomez-Sanchez C, Piper M, Lentz R. Prepectoral Breast Reconstruction in the Setting of Postmastectomy Radiation Therapy: An Assessment of Clinical Outcomes and Benefits. Plast Reconstr Surg. 2019 Jan;143(1):10-20. doi: 10.1097/PRS.0000000000005140. PMID 30589770
- [Result] Garza RM, Paik KJ, Chung MT, Duscher D, Gurtner GC, Longaker MT, Wan DC. Studies in fat grafting: Part III. Fat grafting irradiated tissue--improved skin quality and decreased fat graft retention. Plast Reconstr Surg. 2014 Aug;134(2):249-257. doi: 10.1097/PRS.0000000000000326. PMID 25068325
- [Result] Cano SJ, Klassen AF, Scott AM, Cordeiro PG, Pusic AL. The BREAST-Q: further validation in independent clinical samples. Plast Reconstr Surg. 2012 Feb;129(2):293-302. doi: 10.1097/PRS.0b013e31823aec6b. PMID 22286412
- [Result] Voineskos SH, Nelson JA, Klassen AF, Pusic AL. Measuring Patient-Reported Outcomes: Key Metrics in Reconstructive Surgery. Annu Rev Med. 2018 Jan 29;69:467-479. doi: 10.1146/annurev-med-060116-022831. PMID 29414263